CLINICAL TRIAL: NCT01039402
Title: Connection Between GP's Estimation of Cardiovascular Risk and Theoretical Calculation in France
Brief Title: Connection Between General Practitioner's (GP's) Estimation of Cardiovascular Risk and Theoretical Calculation in France
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: MC MD, AstraZeneca
Other Study IDs: NIS-CFR-DUM-2009/3
Record Dates: First submitted 2009-12-24; First posted 2009-12-25 (Estimated); Last update posted 2010-09-16 (Estimated); Status verified 2010-09

CONDITIONS: Cardiovascular Risk
Keywords: cardiovascular risk; France; Observational, descriptive study

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 1: Adults ≥ 50 years old

SUMMARY:
The purpose of this study is to evaluate connection between GP's estimation of cardiovascular risk and theoretical calculation.

ELIGIBILITY:
Inclusion Criteria:

* Adults 50 years old and over, visiting their GPs

Min Age: 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care
Sampling Method: Probability Sample
Enrollment: 13502 (Estimated)
Dates: Start 2009-12; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
To evaluate connection between GP's estimation of cardiovascular risk and theoretical calculation (according to guidelines and validated scales (such as risk score profile in the Framingham Heart study or the SCORE risk estimation)) | At the end of the study

SECONDARY OUTCOMES:
To estimate the number of cardiovascular risk patients, that have not been identified | At the end of the study
To characterize those patients according to their theoretical cardiovascular risk (high, medium, low) | At the end of the study
to reveal GP's estimation of cardiovascular risk is especially driven by LDL | At the end of the study

CONTACTS AND LOCATIONS:
Overall Officials: Pr Eric BRUCKERT, Study Chair — APHP Paris - France, Hôpital La Pitié-Salpétriêre; Mrs Geneviève BONNELYE, Principal Investigator — KantarHealth - France
Locations (275):
- France (275):
  - Research Site, Ajaccio
  - Research Site, Ancenis
  - Research Site, Andernos-les-Bains
  - Research Site, Andlau
  - Research Site, Andrézieux-Bouthéon
  - Research Site, Angoulême
  - Research Site, Annecy
  - Research Site, Annezin
  - Research Site, Antibes
  - Research Site, Antony
  - Research Site, Arcey
  - Research Site, Arches
  - Research Site, Argences
  - Research Site, Argenteuil
  - Research Site, Arras
  - Research Site, Aubigny-en-Artois
  - Research Site, Aujargues
  - Research Site, Auriol
  - Research Site, Avignon
  - Research Site, Avoine
  - Research Site, Baixas
  - Research Site, Balma
  - Research Site, Banon
  - Research Site, Baumont Les Valence
  - Research Site, Beaumont-sur-Oise
  - Research Site, Belfort
  - Research Site, Belleville
  - Research Site, Benest
  - Research Site, Bergbinten
  - Research Site, Bergerac
  - Research Site, Bersée
  - Research Site, Besançon
  - Research Site, Bessancourt
  - Research Site, Bethoncourt
  - Research Site, Bezanes
  - Research Site, Bétaille
  - Research Site, Béziers
  - Research Site, Biarritz
  - Research Site, Bléré
  - Research Site, Blois
  - Research Site, Bondues
  - Research Site, Bonnieux
  - Research Site, Bordeaux
  - Research Site, Bosmie
  - Research Site, Boulogne-Billancourt
  - Research Site, Bourbriac
  - Research Site, Bourg-de-Thizy
  - Research Site, Brebières
  - Research Site, Brest
  - Research Site, Brivé
  - Research Site, Brunoy
  - Research Site, Buc
  - Research Site, Bugeat
  - Research Site, Cachan
  - Research Site, Caluire-et-Cuire
  - Research Site, Camblain-lAbbé
  - Research Site, Cannes
  - Research Site, Carpentras
  - Research Site, Carquefou
  - Research Site, Carvin
  - Research Site, Chamonix
  - Research Site, Champagnole
  - Research Site, Chaumont
  - Research Site, Châlons-en-Champagne
  - Research Site, Cherbourg
  - Research Site, Chevannes
  - Research Site, Chinon
  - Research Site, Clermont-Ferrand
  - Research Site, Collioure
  - Research Site, Colombey-les-Belles
  - Research Site, Couëron
  - Research Site, Courbevoie
  - Research Site, Courpière
  - Research Site, Coutiches
  - Research Site, Crach
  - Research Site, Croissy-sur-Seine
  - Research Site, Cugnaux
  - Research Site, Dambach-la-Ville
  - Research Site, Devecey
  - Research Site, Digne-les-Bains
  - Research Site, Dijon
  - Research Site, Dole
  - Research Site, Donville-les-Bains
  - Research Site, Douchy-les-Mines
  - Research Site, Elliant
  - Research Site, Espelette
  - Research Site, Espondeilhan
  - Research Site, Échirolles
  - Research Site, Écully
  - Research Site, Fabrezan
  - Research Site, Fenioux
  - Research Site, Fontenay-sous-Bois
  - Research Site, Fouesnant
  - Research Site, Fougères
  - Research Site, Franconville
  - Research Site, Fréhel
  - Research Site, Fronton
  - Research Site, Gonesse
  - Research Site, Gratentour
  - Research Site, Grenoble
  - Research Site, Guérande
  - Research Site, Hay Les Roses
  - Research Site, Houilles
  - Research Site, Irigny
  - Research Site, Jouy-le-Moutier
  - Research Site, La Courneuve
  - Research Site, La Couronne
  - Research Site, La Londe
  - Research Site, La Motte-Servolex
  - Research Site, La Riche
  - Research Site, Lamagistère
  - Research Site, Lambersart
  - Research Site, Lapugnoy
  - Research Site, Latresne
  - Research Site, Lattes
  - Research Site, Laval
  - Research Site, Le Bourget
  - Research Site, Le Chesnay
  - Research Site, Le Grand-Lemps
  - Research Site, Le Havre
  - Research Site, Le Lude
  - Research Site, Le Port-Marly
  - Research Site, Le Quesnoy
  - Research Site, Le Russey
  - Research Site, Les Pennes-Mirabeau
  - Research Site, Les Pujols
  - Research Site, Les Sables-d'Olonne
  - Research Site, Lherbergement
  - Research Site, Lille
  - Research Site, Limeray
  - Research Site, Limoges
  - Research Site, Longtpont Sur Orge
  - Research Site, Louviers
  - Research Site, Lumbin
  - Research Site, Lyon
  - Research Site, Marcq-en-Barœul
  - Research Site, Mareuil-sur-Lay
  - Research Site, Marignane
  - Research Site, Marles-les-Mines
  - Research Site, Marlesmines
  - Research Site, Marquette Les Lille
  - Research Site, Marseille
  - Research Site, Mauléon-Licharre
  - Research Site, Merville
  - Research Site, Metz
  - Research Site, Méounes-lès-Montrieux
  - Research Site, Méréville
  - Research Site, Monteux
  - Research Site, Montigny-le-Bretonneux
  - Research Site, Montigny-lès-Cormeilles
  - Research Site, Montmain
  - Research Site, Montmorillon
  - Research Site, Montpellier
  - Research Site, Montreuil
  - Research Site, Montrond-le-Château
  - Research Site, Montrouge
  - Research Site, Morcenx
  - Research Site, Moreuil
  - Research Site, Mourenx
  - Research Site, Mouvaux
  - Research Site, Nancy
  - Research Site, Nantes
  - Research Site, Narbonne
  - Research Site, Neuilly-Plaisance
  - Research Site, Neuville-en-Ferrain
  - Research Site, Néré
  - Research Site, Nice
  - Research Site, Nieuil-l'Espoir
  - Research Site, Nîmes
  - Research Site, Norges Le Bas
  - Research Site, Noyon
  - Research Site, Oberhausbergen
  - Research Site, Oignies
  - Research Site, Orléans
  - Research Site, Paris
  - Research Site, Pessac
  - Research Site, Peyruis
  - Research Site, Périgueux
  - Research Site, Pérols
  - Research Site, Pierrefitte-sur-Sauldre
  - Research Site, Plabennec
  - Research Site, Pleubian
  - Research Site, Pocé-sur-Cisse
  - Research Site, Poitiers
  - Research Site, Pompey
  - Research Site, Pont Labbe Darnoult
  - Research Site, Pont-Évêque
  - Research Site, Portet-sur-Garonne
  - Research Site, Pouilley-les-Vignes
  - Research Site, Prey
  - Research Site, Privas
  - Research Site, Provins
  - Research Site, Puyricard
  - Research Site, Reims
  - Research Site, Rennes
  - Research Site, Riedishiem
  - Research Site, Rodilhan
  - Research Site, Romainville
  - Research Site, Rosiers Degletons
  - Research Site, Roubaix
  - Research Site, Rousset
  - Research Site, Royan
  - Research Site, Rueil-Malmaison
  - Research Site, Rugles
  - Research Site, Sainghin-en-Mélantois
  - Research Site, Saint Gervais Dauvergne
  - Research Site, Saint Maurice Les Chatauneuf
  - Research Site, Saint-Aigulin
  - Research Site, Saint-Amant-de-Boixe
  - Research Site, Saint-Apollinaire
  - Research Site, Saint-Avold
  - Research Site, Saint-Brieuc
  - Research Site, Saint-Etienne
  - Research Site, Saint-Étienne-les-Orgues
  - Research Site, Saint-Germain-de-la-Coudre
  - Research Site, Saint-Germain-en-Laye
  - Research Site, Saint-Jean-Pied-de-Port
  - Research Site, Saint-Léger-des-Bois
  - Research Site, Saint-Lô
  - Research Site, Saint-martin Dauxigny
  - Research Site, Saint-Michel
  - Research Site, Saint-Nazaire
  - Research Site, Saint-Paul-en-Jarez
  - Research Site, Saint-Prest
  - Research Site, Saint-Prouant
  - Research Site, Saint-Rémy-de-Provence
  - Research Site, Saint-valier
  - Research Site, Sainte-Foy-de-Peyrolières
  - Research Site, Salomé
  - Research Site, Salouël
  - Research Site, Schiltigheim
  - Research Site, Segonzac
  - Research Site, Sète
  - Research Site, Sélestat
  - Research Site, Simiane-Collongue
  - Research Site, Soissons
  - Research Site, Sonchamp
  - Research Site, Strasbourg
  - Research Site, Suippes
  - Research Site, Théoule-sur-Mer
  - Research Site, Thiviers
  - Research Site, Thorigné-Fouillard
  - Research Site, Thouaré-sur-Loire
  - Research Site, Thun-Saint-Amand
  - Research Site, Tionville
  - Research Site, Toulon
  - Research Site, Toulouse
  - Research Site, Tourcoing
  - Research Site, Tours
  - Research Site, Toussieu
  - Research Site, Uchaud
  - Research Site, Ussel
  - Research Site, Uxem
  - Research Site, Valence Dalbigeois
  - Research Site, Vandœuvre-lès-Nancy
  - Research Site, Vanves
  - Research Site, Vaugneray
  - Research Site, Vennecy
  - Research Site, Verneuil-sur-Avre
  - Research Site, Verson
  - Research Site, Veynes
  - Research Site, Vezins
  - Research Site, Villejuif
  - Research Site, Villeneuve Dascq
  - Research Site, Villeneuve-Loubet
  - Research Site, Villennes-sur-Seine
  - Research Site, Villers-lès-Nancy
  - Research Site, Villeurbanne
  - Research Site, Vincennes
  - Research Site, Visan
  - Research Site, Voiron
  - Research Site, Wasquehal
  - Research Site, Wasselonne
  - Research Site, Witry-lès-Reims
  - Research Site, Wœrth